CLINICAL TRIAL: NCT01361685
Title: Attain Ability® Family Left Ventricular Lead Chronic Performance Study
Brief Title: Model 4396 Left Ventricular (LV) Lead Chronic Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4396 Chronic Performance
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lead survivability will be summarized.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate long-term performance of the 4396 LV Lead. This evaluation is based on the number of lead-related complications occurring during the study compared to the number of leads enrolled in the study. The leads will be followed for 5 years after implant. This study is required by FDA as a condition of approval of the Model 4396 LV Lead. This study is conducted within Medtronic's post-market surveillance platform.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and do not meet any of the following exclusion criteria are eligible for enrollment.

Inclusion Criteria

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive an Attain Ability Model 4396 LV lead
* Patient within 30 day post implant enrollment window

Exclusion Criteria

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with a 4396 LV Lead within 30 days. All subjects must meet Inclusion criteria and none of the Exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2011-05; Primary Completion 2020-03-02 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Model 4396 LV Lead-related complication rate | 5 years

SECONDARY OUTCOMES:
Types of lead-related adverse device effects | 5 years
Percent of subjects with changes in electrode programming | 5 years
Number of fractures with and without loss of function | 5 years
Bipolar electrical performance at 1 year | 1 year
Bipolar pacing impedance | 1 year
Bipolar pacing capture threshold | 1 year

CONTACTS AND LOCATIONS:
Locations (52):
- United States (48):
  - Southwest EP Clinic, Gilbert, Arizona
  - Saint Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - COR Healthcare, Torrance, California
  - Cardiovascular Consultants Medical Group, Van Nuys, California
  - Colorado Heart and Vascular, PC, Lakewood, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Southern Maryland Hospital Center, Washington D.C., District of Columbia
  - Bradenton Cardiology, Bradenton, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - Indiana University Health - Methodist Research Institute, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Louisville Cardiology Group, Louisville, Kentucky
  - Cenla Heart Specialists, Alexandria, Louisiana
  - Our Lady of the Lake Office of Research, Baton Rouge, Louisiana
  - Michigan Heart, Ypsilanti, Michigan
  - Metropolitan Cardiology Consultants PA, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - HealthCare Partners Medical Group, Saint Louis Park, Minnesota
  - Saint Lukes Health System, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Patients First Health Care LLC, Washington, Missouri
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - New York-Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Central New York Cardiology, Utica, New York
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - The Christ Hospital Health Network, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Lehigh Valley Health Network, Bethlehem, Pennsylvania
  - Medicor Associates, Erie, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - STAR Clinical Trials, San Antonio, Texas
  - EP Heart LLC, The Woodlands, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Canada (3):
  - Queen's University & Kingston General Hospital, Kingston, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM) Hopital Hotel-Dieu, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec
- Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg, Germany